CLINICAL TRIAL: NCT05210036
Title: Comparison of The Effectiveness of High-intensity Laser and Ultrasound Therapies in Adhesive Capsulitis: A Randomized Controlled Study
Brief Title: HILT and US Therapies in Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Bilal Uysal, Assistant Professor, Balikesir University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Physical Medicine
Record Dates: First submitted 2021-12-30; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Adhesive Capsulitis of Shoulder
Keywords: Frozen Shoulder, Ultrasound, High-Intensity Laser Therapy
MeSH Terms: conditions — Bursitis | interventions — Ultrasonic Therapy; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound Therapy (Active Comparator): The patients in group 1 received therapeutic US with BTL-4710 ultrasound device.
  The therapeutic US was administered at the frequency of 3 megahertz, intensity of 1.5 w/cm2 and an area of 25 cm2 for 5 minutes in the continue mode.
  The procedure of therapeutic US was performed by a physiotherapist experienced in using the device for 15 sessions in total 5 times a week for 3 weeks.
  Interventions: Device: Ultrasound Therapy (US)
- High-Intensity Laser Therapy (Active Comparator): The patients in group 2 received HILT with BTL-6000 high-intensity laser device.
  The therapy consisted of 2 stages in each session.
  * The first stage was performed in analgesic mode for analgesic effect at the frequency of 25 Hz, in the wavelength of 1064 nm, the power of 8 watt, the dose of 12 j/cm2, the area of 25 cm2, and 300 j in total for 2 minutes and 30 seconds.
  * The second stage was performed in bio-stimulating mode for biostimulation effect in the wavelength of 1064 nm, the power of 7 watt, the dose of 100 j/cm2, the area of 25 cm2, and 2500 j in total for 5 minutes and 57 seconds.
  The total length of administration was approximately 8.5 minutes for each stage.
  The procedure of the therapy was performed by a physiotherapist experienced in using the device for 9 sessions in total 3 times a week for 3 weeks.
  Interventions: Device: High-Intensity Laser Therapy (HILT)

INTERVENTIONS:
Device: Ultrasound Therapy (US) — All the patients included in the study received a total of 15 sessions of physical therapy program 5 times a week for 3 weeks.
  Physical Therapy Program;
  * Hot Pack at 60 degrees Celsius for 20 minutes
  * TENS at 80 Hz for 20 minutes
  * Therapeutic exercise program (3 sets of 10 reps with 3-minute intervals between the sets) consisting of active-assisted ROM, passive stretching and Codman exercises for their shoulder joint for 30 minutes in accompany with a physiotherapist.
  Other Names: Transcutaneous Electrical Nerve Stimulation (TENS); Hot Pack; Therapeutic Exercise Program
  Arms: Ultrasound Therapy
Device: High-Intensity Laser Therapy (HILT) — All the patients included in the study received a total of 15 sessions of physical therapy program 5 times a week for 3 weeks.
  Physical Therapy Program;
  * Hot Pack at 60 degrees Celsius for 20 minutes
  * TENS at 80 Hz for 20 minutes
  * Therapeutic exercise program (3 sets of 10 reps with 3-minute intervals between the sets) consisting of active-assisted ROM, passive stretching and Codman exercises for their shoulder joint for 30 minutes in accompany with a physiotherapist.
  Other Names: Transcutaneous Electrical Nerve Stimulation (TENS); Hot Pack; Therapeutic Exercise Program
  Arms: High-Intensity Laser Therapy

SUMMARY:
Background: Adhesive capsulitis (AC) is a common musculoskeletal disease characterized by pain and limitation of movement in the shoulders of patients.

Purpose: This study aimed to assess the effectiveness of short- and long-term therapeutic ultrasound (US) and high-intensity laser therapy (HILT) in the treatment of AC.

Methods: A total of 60 patients with AC were randomized into two groups. Group I received US (15 sessions in total) and Group II received HILT (9 sessions in total) for 3 weeks. In addition, all the patients received 15 sessions of physical therapy programs (hot pack, TENS and therapeutic exercises). Assessments were made using VAS-Pain, Shoulder Pain and Disability Index (SPADI) and range of motion (ROM) with goniometer before and at the end of the treatment and in the posttreatment 1st and 6th months.

DETAILED DESCRIPTION:
INTRODUCTION AC is a common musculoskeletal disease characterized with pain on the patients' shoulder, movement restriction and insufficiency in daily life activities [1]. The prevalence of AC is between 2-5% in general population and higher between the ages of 40 and 60 and among women [2].

The aim in the treatment of AC is to relieve pain and increase the joint range of motion (ROM) and functioning [5]. The treatment of AC remains controversial because the level of evidence for various treatments is limited [6]. Controlled prospective studies are difficult to design and perform because of controversies in the definition, classification, diagnosis and stages of AC [6]. Many different treatment methods such as medical treatment, physical therapy, exercises, intraarticular steroid injections, suprascapular nerve block, manipulation under anesthesia, and surgical interventions are used in the treatment of AC [7]. Although many different treatment methods are used in the treatment of AC there is no consensus on the standard treatment method. Positive effects of physical therapy practices on AC in the short and long term have been revealed [8].

Among physical therapy practices, superficial and deep heating agents (infrared radiation, hot pack, shortwave diathermy, low-density laser therapy, HILT and US, etc.), electrotherapy modalities (Transcutaneous Electrical Nerve Stimulation (TENS), diadinamic current, galvanic current, etc.) and exercises are used alone or in combination in the treatment of AC [9]. Therapeutic US is often used in physical therapy practices in the treatment of AC and the interest in HILT has recently been increasing as well [10].

This study aimed to investigate whether there was a difference between therapeutic US and HILT in terms of the short-term and long-term effects on pain, ROM and functional condition in the treatment of AC.

METHODS The study was designed as a prospective, randomized, controlled, and single-blind study. A total of 60 patients who were admitted to the physical therapy and rehabilitation outpatient clinic with pain and movement restriction in their shoulder and who signed the patient information consent form were included in the study.

A total of 60 patients who met the inclusion criteria of the study were divided into 2 groups (30 patients in each group) with simple randomization method by using a table of random numbers created on the computer. The researchers who made the assessment measurements were unaware of which patient was in which group. Statistical analysis of the results was performed by a biostatistician who had no information about the therapies the patient groups received.

All the patients included in the study received a total of 15 sessions of physical therapy program 5 times a week for 3 weeks. All the patients received hot pack at 60oC for 20 minutes and conventional TENS at 80 Hz for 20 minutes for their involved shoulder. In addition to these therapies, the patients in group 1 received US and those in group 2 received HILT. After physical therapy, all the participants received therapeutic exercise program (3 sets of 10 reps with 3-minute intervals between the sets) consisting of active-assisted ROM, passive stretching and Codman exercises for their shoulder joint for 30 minutes in accompany with a physiotherapist. Interventions for groups; Grup 1 (US) = US + Hot Pack + TENS + Therapeutic Exercise Program Grup 2 (HILT) = HILT + Hot Pack + TENS + Therapeutic Exercise Program The patients were assessed with the measurements of visual analogue scale (VAS)-pain, Shoulder Pain and Disability Index (SPADI) and ROM with goniometer before and at the end of the treatment and in the posttreatment 1st and 6th months.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with primary (idiopathic) AC,
* Pain and movement restriction in his or her shoulder for at least 3 months,
* Restriction of passive external rotation in the involved shoulder restricted with less than 50% of the contralateral shoulder,
* Normal radiography findings

Exclusion Criteria:

* Both shoulders were involved,
* Other shoulder pathologies (glenohumeral osteoarthritis, calcific tendinitis, rotator cuff tear, etc.),
* Cervical radiculopathy,
* Brachial plexus lesion,
* Neuromuscular disorders,
* Inflammatory rheumatic disorders,
* Malignancy,
* Acute trauma,
* Patients who had fracture affecting the involved shoulder joint, patients who underwent a surgical intervention, patients who underwent intraarticular injection for the involved shoulder within the last 6 months,
* Patients who received physical therapy for the glenohumeral joint within the last 1 year, and
* Photoallergy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11-15 (Actual); Primary Completion 2016-05-15 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS)-pain, | "at the end of the treatment, week 3", "at the end of the treatment, month 1" "at the end of the treatment, month 6"
  Detection of improvements in VAS-pain,
Shoulder Pain and Disability Index (SPADI) | "at the end of the treatment, week 3", "at the end of the treatment, month 1" "at the end of the treatment, month 6"
  Detection of improvements in SPADI
Joint range of motion (ROM) | "at the end of the treatment, week 3", "at the end of the treatment, month 1" "at the end of the treatment, month 6"
  Detection of improvements in joint range of motion (ROM) with goniometer

IPD SHARING:
Plan to Share IPD: No